CLINICAL TRIAL: NCT04606693
Title: Value of Screening and Treatment of Sleep Apnea-Hypopnea Syndrome in the Management of Atrial Fibrillation Ablation Candidates
Brief Title: Value of Screening and Treatment of SAHS in the Management of AF Ablation Candidates
Acronym: SLEEP-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Nicasio Perez Castellano, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20/023-E
Record Dates: First submitted 2020-01-16; First posted 2020-10-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation Paroxysmal; Atrial Fibrillation, Persistent; Apnea Syndrome; Hypopnea Syndrome
Keywords: Atrial Fibrillation; Apnea; Hypopnea; SAHS
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with negative diagnosis of SAHS (No Intervention): Patients with low risk or negative diagnosis of SAHS will follow conventional management of their AF, according to the usual criteria of the Arrhythmia Unit
- Patients with positive diagnosis of SAHS (Other): Patients with intermediate or high risk of SAHS and positive diagnosis
  Interventions: Other: Treatment of SAHS

INTERVENTIONS:
Other: Treatment of SAHS — Patients diagnosed with SAHS will be treated in the Pneumology Service according to usual practice (dietary hygienic measures, CPAP, etc.).
  Arms: Patients with positive diagnosis of SAHS

SUMMARY:
The present prospective cohort study (not randomized) analyses the value of screening and treatment of SAHS in the management of patients with AF refractory to antiarrhythmics drugs, potentially candidates for ablation.

Patients at low risk of suffering from SAHS will follow conventional management of their AF, according to the usual criteria of the Arrhythmia Unit. Patients with high or intermediate risk of SAHS, will undergo respiratory polygraphy. If the result is positive, they will be treated as standard for this syndrome and their heart rate will be monitored for 3 months. After this, the patient's arrhythmic load will be reevaluated differentiating patients into two groups, those that must be ablated from those that have improved their condition and the clinical criteria is no longer ablation but follow-up.

DETAILED DESCRIPTION:
All patients who meet all the inclusion criteria and none of the exclusion will have a Stop-Bang questionnaire to define the risk of having a SAHS The assessment of results classifies people at high, intermediate or low risk of SAHS. Low-risk patients will follow conventional management according to the usual criteria of the Arrhythmia Unit.

Patients with high or intermediate-risk will be given a Kardia© recorder and they will be instructed to obtain records of their cardiac rhythm every 5 days (at any time) and whenever the symptoms are suggestived of arrhythmia. This allows estimating arrhythmic load baseline in these patients.

They will also will be given a 7-channel home respiratory polygraphy (with pulse oximetry record, naso-buccal air flow through nasal cannula and thermistor, snoring, thoracoabdominal movements and electrocardiogram). The day after conducting the home polygraphic record, the patient will be evaluated in the Pneumology Outpatient Department, where risk factors, symptoms and Epworth's sleepiness scale will be assessed, the results of the cardiorespiratory polygraphic record, interpreted by Pneumology Service will be given , and based on the above, the diagnosis of SAHS will be determined.

Those patients diagnosed with SAHS will be treated in the Pneumology Service according to usual practice (dietary hygienic measures, CPAP, etc.).

During all this time, patients will continue using their rhythm recorders as previously. The overall effect of SAHS treatment on AF recurrences (comparison of arrhythmic load in the previous 3 months with that of the 3 months post-treatment) will be evaluated.

After 3 months of starting the treatment, a follow-up respiratory polygraphy will be carried out, where the relationship between the changes in AHI and desaturation index as well as changes in arrhythmic load will be evaluated.

Once the follow-up respiratory polygraphy is performed, the indication of AF ablation will be reassessed. Patients who continue with symptomatic recurrences of AF refractory to antiarrhythmics will undergo ablation.

It will be analyzed that proportion of patients initially candidates for ablation cease to fulfill conditions for this by a better control of recurrences and "leave the waiting list". Likewise, the results of the ablation of the cohort of patients diagnosed with SAHS and the moderate or high-risk cohort of SAHS, but with negative polygraphy and diagnosis, will be compared.

The arrhythmic load after AF ablation will be analysed, during the blinding period (3 months post-ablation) and one year after the ablation. Patients will continue their SAHS treatment according to the usual practice of the Pneumology Service.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent atrial fibrillation
* Recurrent atrial fibrillation despite treatment with at least one class I or III antiarrhythmic
* No previous diagnosis of apnea-hypopnea syndrome

Exclusion Criteria:

* Patients <18 years
* Pregnant women
* Doubts about the patient's ability to perform a home respiratory polygraphy
* Doubts about the patient's ability to acquire rhythm records with the Kardia system (smartphone required)
* Unavailability for follow-up at our center for at least 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Arrhythmic load | Six months
  Rate of time in FA measured with Kardia © recorder

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain